CLINICAL TRIAL: NCT03258788
Title: A Translational Study Investigating PD-L1 Expression After Radiotherapy for Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Translational Study Investigating PD-L1 Expression After Radiotherapy for Non-small Cell Lung Cancer
Acronym: PD-RAD
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CFTSp095, 14_DOG07_183
Record Dates: First submitted 2017-08-10; First posted 2017-08-23 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Original diagnostic tumour blocks will be returned at the end of the study. New biopsy and blood samples taken may be used in future research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Small Cell Lung Cancer: Participants with NSCLC not suitable for concurrent CTRT, being treated with standard radiotherapy (radical or palliative). All participants will be required to undergo a post radiotherapy course biopsy and will have blood samples taken.
  Interventions: Procedure: Biopsy and blood samples

INTERVENTIONS:
Procedure: Biopsy and blood samples — Archival tumour biopsies will be analysed for baseline PD-L1 expression. Some participants will have a biopsy before radiotherapy if the archival biopsy is not suitable.
  Participants will be required to undergo an additional mandatory biopsy of the irradiated site during the second week. Patients must have completed at least 1 week of the planned treatment before taking the biopsy.
  Participants will also be asked for consent to donate 50ml blood pre biopsy (at baseline and week 2) and at the end of radiotherapy; as well as 10ml blood before #2 radiotherapy and weekly throughout treatment.

SUMMARY:
Participants with Non-Small Cell Lung Cancer (NSCLC), Performance Status (PS) 0-2, not suitable for concurrent Chemo-Radiotherapy (CTRT), will be treated with standard radiotherapy (radical or palliative). Archival tumour biopsies will be analysed for baseline Programmed Death Ligand 1 (PD-L1) expression. Some participants will have a biopsy before radiotherapy if the archive biopsy is not suitable. Participants will be required to undergo an additional mandatory biopsy of the irradiated site during the second week of radiotherapy.

DETAILED DESCRIPTION:
The purpose of this prospective, multicentre, non-randomised translational study is to provide proof of feasibility of achieving paired biopsies for PD-L1 assessment in patients with NSCLC treated with palliative or radical radiotherapy. This is a non-CTIMP study.

All participants will have a minimum of 1 mandatory biopsy (during radiotherapy [irradiated site]) and the potential to have a pre-treatment biopsy if archival biopsy does not meet the suitability criteria.

Participants will have up to a maximum of 2 additional optional biopsies (during radiotherapy [within the RT field e.g supraclavicular fossa node], [outside RT field e.g. skin met]).

Blood samples will also be taken on study at specified time points for immune monitoring (exploratory endpoints).

The study will be carried out in two stages as follows:

Stage 1:

Following the enrolment of the first 15 evaluable participants, an interim analysis will take place by the Trial Steering Committee (TSC). The TSC will make a recommendation on whether recruitment should continue to the Trial Management Group (TMG).

Stage 2:

A further 15 evaluable participants will be recruited onto the study to achieve a total of 30 evaluable participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC
* Diagnostic/pre-treatment biopsy suitable for PD-L1 analysis*
* Tumour judged inoperable by a lung MDT
* Tumour that is accessible to core biopsy
* Age 18 and over, no upper age limit
* Performance status (PS) - ECOG 0-2
* Participant considered suitable for radiotherapy (palliative or radical) or sequential chemo-radiotherapy
* Before participant registration, written informed consent must be given according to GCP and national regulations

  * Pre-treatment biopsy must be from gross tumour volume within planned radiation field, and must also:

    * have been formalin fixed for >12h and ≤24h
    * have tumour tissue and morphology confirmed by H&E staining
    * contain sufficient tumour cells (>100) to determine PD-L1 status

Exclusion Criteria:

* Participant suitable for standard concurrent CTRT
* Participant deemed unsuitable for repeat biopsies in the opinion of the treating oncologist
* Participant known to have an EGFR mutation or an ALK rearrangement
* Intercurrent or history of hepatitis B, C or human immunodeficiency virus infection, if known
* Participants who have received more than 1 line of chemotherapy prior to radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Achieving paired biopsies for PD-L1 assessment in 21 of the 30 evaluable participants | Up to 6.5 weeks from start of radiotherapy

SECONDARY OUTCOMES:
Suitability of pre and during radiotherapy biopsy for PD-L1 testing | Up to 6.5 weeks from start of radiotherapy

OTHER OUTCOMES:
Change in PD-L1 expression level during treatment | Up to 6.5 weeks from start of radiotherapy
Difference in PD-L1 expression level in 'out of radiotherapy field' sites compared with irradiated sites | Up to 6.5 weeks from start of radiotherapy
Immune monitoring of primary tumour and peripheral blood mononuclear cells | Up to 6.5 weeks from start of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Illidge, Study Chair — The Christie NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - St. James's Univerisity Hospital, Leeds
  - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- See also: End of Trial Report - HRA — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/pd-rad/
- See also: University of Manchester - Website — https://research.manchester.ac.uk/en/publications/pd-rad-a-translational-study-investigating-pd-l1-expression-after